CLINICAL TRIAL: NCT03004287
Title: 2015-12: A Phase II Study Exploring the Use of Early and Late Consolidation/Maintenance With Anti-CD38 (Protein) Monoclonal Antibody to Improve Progression Free Survival in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: 2015-12: A Study Exploring the Use of Early and Late Consolidation/Maintenance Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206241
Record Dates: First submitted 2016-12-19; First posted 2016-12-28 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Thalidomide; Dexamethasone; Calcium Dobesilate; daratumumab; Cisplatin; Doxorubicin; Cyclophosphamide; Etoposide; Melphalan; Lenalidomide; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Treatment (Experimental): Induction Chemotherapy: Carfilzomib, Thalidomide, Dexamethasone, Daratumumab , CisPlatin, Adriamycin, Cyclophosphamide and Etoposide (KTD-Dara-PACE).
  Autologous Stem Cell Transplant (ASCT) 1: Melphalan, Dexamethasone, ASCT.
  Immunological Consolidation 1: Daratumumab.
  Consolidation 1: Daratumumab, Carfilzomib, Dexamethasone (Dara-KD).
  ASCT 2 (optional): Melphalan, Dexamethasone, ASCT.
  Immunological Consolidation 2: Daratumumab.
  Maintenance: Dara-KD alternating with Daratumumab, lenalidomide, and Dexamethasone (Dara-RD) in 3-month blocks.
  Bortezomib may be substituted for carfilzomib throughout the regimen at the discretion of the treating physician.
  Interventions: Drug: Carfilzomib; Drug: Thalidomide; Drug: Dexamethasone; Drug: Daratumumab; Drug: Cisplatin; Drug: Adriamycin; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Melphalan; Procedure: ASCT; Drug: Lenalidomide; Drug: Bortezomib

INTERVENTIONS:
Drug: Carfilzomib — Given by vein: days 1 and 2 of Induction; days 1, 8, 15, and 22 of Consolidation 1; and days 1, 8, 15, and 22 of alternating 3-month blocks during Maintenance.
  Other Names: Kyprolis
Drug: Thalidomide — Given by mouth at bedtime: days 1-4 of Induction
  Other Names: Thalomid
Drug: Dexamethasone — Given by mouth or by vein: days 1-4 of Induction; days -4 - -1 of Transplant(s); and days 1, 8, 15, and 22 of every cycle during Maintenance
  Other Names: Baycadron
Drug: Daratumumab — Given by vein: day -1 of induction; days 1 and 8 of Immunological Consolidations; and day 1 of each Maintenance cycle
  Other Names: Darzalex
Drug: Cisplatin — Given by vein: days 1-4 (continuous infusion) of Induction
  Other Names: Platinol
Drug: Adriamycin — Given by vein: days 1-4 (continuous infusion) of Induction
  Other Names: Doxorubicin
Drug: Cyclophosphamide — Given by vein: days 1-4 (continuous infusion) of Induction
  Other Names: Cytoxan
Drug: Etoposide — Given by vein: days 1-4 (continuous infusion) of Induction
  Other Names: Eposin
Drug: Melphalan — Given by vein: days -4 - -1 of Transplant(s)
Procedure: ASCT — day 0 of Transplant(s)
Drug: Lenalidomide — Given by mouth: days 1-21 of alternating 3-month blocks during Maintenance
  Other Names: Revlimid
Drug: Bortezomib — Given by vein or subcutaneous injection: may be substituted for carfilzomib throughout the study regimen at the discretion of the treating physician
  Other Names: Velcade

SUMMARY:
This study will assess whether adding one of the newest multiple myeloma therapies, daratumumab, into the Total Therapy approach helps patients live longer with fewer side effects

DETAILED DESCRIPTION:
Past studies conducted at the Myeloma Institute and at other institutions have shown that many patients with high-risk disease (as determined by gene array studies - studies that look at specific genes using special equipment) tend to have shorter remissions (disappearance of signs and symptoms of myeloma) and do not survive as long as participants with low-risk myeloma. The Total Therapy approach to treatment carried out at the Myeloma Institute where multiple chemotherapy agents are given as induction followed by a stem cell transplant, post-transplant consolidation, and maintenance therapy has proven to be the best available treatment strategy. However, the availability of new treatments that work in different ways offers the possibility of improving the effectiveness of Total Therapy treatment while potentially reducing the number of side effects patients' experience. Daratumumab is a human monoclonal antibody or protein drug. It recognizes a specific protein, CD38, which is found at high levels on multiple myeloma cells. An antibody is something that finds and kills foreign objects in your body, in this case, myeloma cells. The other drugs that will be used in the study treatment regimen include carfilzomib or bortezomib, thalidomide, lenalidomide, dexamethasone, cisplatin, adriamycin, cyclophosphamide, etoposide, lenalidomide and dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed active Multiple Myeloma (MM) requiring treatment. Patients with a previous history of smoldering myeloma will be eligible if there is evidence of progressive disease requiring chemotherapy.
* Patients must be either untreated or have not received more than four cycles of systemic MM therapy (e.g. Revlimid Dexamethasone (RD), Bortezomib Revlimid Dexamethasone (VRD). Prior bisphosphonates and localized radiation are allowed.
* Participants must have high-risk disease, as defined by at least one of the following:
* Myeloma Prognostic Risk Signature (MyPRS) risk score ≥ 50.4
* Lactate Dehydrogenase (LDH) ≥ 360 U/L (Rule out hemolysis and infection; contact PI if any doubt.)
* Diagnosis of primary plasma cell leukemia.
* Eastern Cooperative Oncology Group (ECOG) ≤ 2, unless solely due to symptoms of MM-related bone disease.
* Patients must have a platelet count ≥ 50,000/μL, unless lower levels are explained by extensive bone marrow plasmacytosis.
* Patients must be at least 18 years of age and not older than 75 years of age at the time of registration.
* Participants must have a baseline serum creatinine level < 3 mg/dL and baseline Alanine Aminotransferase (ALT) < 3x Upper Limit of Normal (ULN).
* Participants must have an ejection fraction by echocardiogram (ECHO) or Multiple-gated Acquisition Scan (MUGA) scan ≥ 45%
* Patients must have adequate pulmonary function studies > 50% of predicted on mechanical aspects (Forced Expiratory Volume 1 (FEV1), Forced Vital Capacity (FVC) and diffusion capacity (DLCO) > 50% of predicted. If the patient is unable to complete pulmonary function tests due to MM related pain or other conditions, an exception may be granted if the principal investigator documents that the patient is a candidate for high dose therapy.
* Patients must have signed an Institutional Review Board (IRB)-approved informed consent indicating their understanding of the proposed treatment and that the protocol has been approved by the Institutional Review Board (IRB).

Exclusion Criteria:

* No evidence of high-risk disease
* Poorly controlled hypertension, diabetes mellitus, active or uncontrolled hepatitis, or other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
* Patients must not have prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has not received treatment for one year prior to enrollment. Other cancers will only be acceptable if the patient's life expectancy exceeds five years.
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy documented within one week of registration.
* Subjects of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Measure the progression-free survival in patients with high risk multiple myeloma | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Frits van Rhee, MD, Principal Investigator — University of Arkansas for Medical Science-Myeloma Institute
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pawlyn C. High-risk myeloma: a challenge to define and to determine the optimal treatment. Lancet Haematol. 2021 Jan;8(1):e4-e6. doi: 10.1016/S2352-3026(20)30361-6. Epub 2020 Dec 22. No abstract available. PMID 33357481